CLINICAL TRIAL: NCT03858647
Title: Multi-Center Assessment of Electrode Placement and Audiologic Outcomes in Cochlear Implantation With the Advanced Bionics HiFocus L23 Electrode
Brief Title: Electrode Placement and Audiologic Outcomes With the Advanced Bionics HiFocus L23 Electrode
Status: Terminated | Type: Observational
Why Stopped: device under study complication-due to PI departure, study closed and will not reopen
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Robert F. Labadie, Professor, Vanderbilt University Medical Center
Other Study IDs: 181904
Record Dates: First submitted 2019-02-12; First posted 2019-03-01 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sensorineural hearing loss patients post cochlear implant: Patients who have documented sensorineural hearing loss and have received cochlear implantation (per standard of care).

SUMMARY:
The goal of this study is to measure patient performance after cochlear implantation with the Food and Drug Administration (FDA) approved Advanced Bionics HiFocus L23 device.

The specific aims of the project are as follows:

1. To measure implant audiologic performance as defined by speech performance in standard cochlear implant speech test batteries.
2. To determine scalar location after insertion through either intraoperative or postoperative imaging and correlate this with audiologic outcomes.
3. To assess the rates of preservation of residual acoustic hearing and correlate those with scalar location as determined in specific aim 2 and audiologic performance as determined in specific aim 1.
4. To correlate speech outcomes with quality of life measures, as defined by validated questionnaires including the Tinnitus Handicap Index (THI), Speech and Spatial Qualities (SSQ) Questionnaire, and Nijmegen Questionnaire.
5. To evaluate intraoperative ease of insertion from the surgeon's perspective and correlate this with postoperative electrode location and audiologic performance.

DETAILED DESCRIPTION:
Cochlear implants (CI) are biomechanical sense prostheses approved by the FDA for the treatment of sensorineural hearing loss. CI's function by bypassing the absent or dysfunctional cochlear end organs to directly electrically stimulate the spiral ganglion and cochlear nerve. A variety of commercially available FDA-approved implants exist for the treatment of severe to profound deafness. Implants are typically designed in two broad categories: lateral wall electrodes and perimodiolar. Perimodiolar electrodes are precurved electrodes that are designed to hug the center of the cochlea (modiolus) after insertion. Lateral wall electrodes are slim and straight, hugging the lateral wall on insertion.

Recent studies have shown that electrode design and location within the cochlea impact patient performance. Specifically, electrodes located completely within the scala tympani are associated with better outcomes than those that cross over from the scala tympani to the scala vestibuli during insertion. The same study has shown that lateral wall electrodes are less likely than perimodiolar electrodes to have scalar excursion to the scala vestibuli. Location matters with these implants because electrode position completely within the scala tympani is associated with higher rates of preservation of residual hearing. Minimizing cochlear trauma allows for preservation of residual acoustic hearing particularly in low frequencies. While this low frequency hearing is of little benefit independently, when combined with the electrical stimulation from the cochlear implant patients have improved performance.

The HiFocus L23 electrode is manufactured by Advanced Bionics (Valencia, California), and is FDA approved for the treatment of sensorineural hearing loss in adult and pediatric patients. It is designed as a slim and straight lateral wall electrode that can be inserted with low force to minimize intracochlear trauma. While pre-market studies were performed by Advanced Bionics as a part of its approval for use by the FDA, no post-market studies have been performed to assess the audiologic outcomes, electrode location after insertion, and hearing preservation rates when using this electrode. These aims will be accomplished through several means. Audiologic speech performance will be assessed through a standardized clinical/audiometric protocol currently followed by the Vanderbilt University Medical Center cochlear implant team. Electrode location for all participants will be determined using novel software created by Vanderbilt engineering faculty and graduate students that uses computerized tomography (CT) images obtained as a part of practice postoperatively or intraoperatively using an FDA approved Xoran xCAT® device, a portable flat panel volume computerized tomography (fpVCT) machine (Vanderbilt) or regular CT scan at participating institutions as applicable. These images can be registered to existing pre-operative conventional CT scans and used to produce 3-dimensional models of electrode placement within each patient's cochlea. This software is investigational and used in other research studies for the same purpose.

The extent to which the electrode remains in the desired location (scala tympani) will then be correlated with audiologic outcomes as obtained above. Residual hearing rates and quality of life measures will be obtained as a part of audiologic testing.

If a fine resolution, high quality conventional head CT has been previously obtained, or is obtained as part of routine care this scan may be used in place of the fpVCT or in addition to the fpVCT scan. The option of having a conventional head CT performed in radiology for research purposes in place of the fpVCT head CT scan will also be available.

Surgeons will complete surveys after each case concludes to evaluate the ease of insertion and will record the insertion via standard recording techniques in the operating room that are available for any microscopic case. These videos for all surgeries will be blinded and reviewed at Vanderbilt for ease and speed of insertion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and above.
* Sensorineural hearing loss meeting criteria for cochlear implants, assessed no greater than three months prior to cochlear implant surgery
* Patient schedule to undergo CI surgery using Advanced Bionics SlimJ/L23 device.
* Ability to undergo adequate audiology follow-up or planned follow up for those participants undergoing scanning in the OR.
* Competent in decision making process and able to read and sign a written informed consent form.
* English language proficiency.
* If the patient has already had a fine resolution CT or a fpVCT of the head (more than likely as a participant of another research study) the scan will not be repeated, the images from the previous scan will be used for the purposes of this study.
* If the patient has undergone a conventional CT scan of the head after cochlear implantation as part of their routine care, this scan may be used in place of the research scan or in addition to the research scan.

Exclusion Criteria:

* Patients who weigh over 300 lbs (when Xoran xCAT headboard is being used). Otherwise, weight is not exclusionary.
* Females who are pregnant. All females of child-bearing age in the study will undergo a pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All clinically confirmed sensorineural hearing loss patients who meet criteria for cochlear implantation using the Advanced Bionics HiFocus L23 electrode are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment Effectiveness-Consonant Nucleus Consonant (CNC) word test | 2 years
  Audiologic speech performance as measured by CNC word recognition. CNC word tests consist of a 50 word list. Subjects repeat as much of each word as possible. Word scores will be calculated as percent correct at baseline through 24 months and reported as percentage points improved.
Treatment Effectiveness-AzBio sentence test | 2 years
  Audiologic speech performance as measured by AzBio sentence recognition. AzBio consists of 20 sentence list spoken by different talkers (two male, two female). Subjects repeat as much of each sentence as possible. Each word correctly repeated counts towards the overall score, reported as an overall percentage correct at baseline through 24 months.
Treatment Effectiveness-Air-conduction thresholds | 2 years
  Audiologic speech performance as measured by air-conduction thresholds. Threshold values will be obtained for 125, 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000, and 8000 Hz using insert earphones. Post-operative hearing thresholds will be compared to pre-operative hearing thresholds to assess amount of residual hearing. Greater post-operative thresholds is associated with poorer hearing preservation.

SECONDARY OUTCOMES:
Treatment Effectiveness | 2 years
  Determine scalar location after electrode insertion using intraoperative or postoperative imaging to then correlate imaging with audiologic outcomes as collected above.
Treatment Effectiveness - Audiologic outcomes | 2 years
  Percentage of residual acoustic hearing for each subject as measured by the audiologic outcomes as collected above.
QOL Tinnitus Handicap Index (THI) | 2 years
  Patient quality of life assessment: tinnitus compared post-implant to pre-implant. The sum of all responses to 25 questions is the THI score, with a range from 0-100. The higher the score, the more handicap the subject has due to tinnitus.
QOL Speech, Spatial and Qualities of Hearing scale (SSQ 12) | 2 years
  Patient quality of life assessment: hearing and listening ability compared post implant to pre-implant. The SSQ 12 survey uses a visual analog rating scale from 0-10 over three listening domains: speech understanding in various listening conditions; spatial hearing associated with distance, movement, and direction; and the overall quality of speech including clarity and naturalness of sound. The higher the score, the better speech understanding, spatial hearing, and sound quality a subject has.
QOL Nijmegen | 2 years
  Patient quality of life assessment: hearing ability scores compared post-implant to pre-implant. The Nijmegen is a 60 question survey covering three general domains: physical, psychological, and social functioning. Subjects rate each question on a scale of how often they can hear an event as noted. The subdomain mean score for each subject is derived by assigning values to survey items as follows: 1 = 0, 2 = 25, 3 = 50, 4 = 75, and 5 = 100 and then calculating the quantitative mean scores across the subdomains.
Evaluation of intraoperative ease of electrode insertion as assessed by surgeon. | 2 years
  Surgeon survey

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Rivas, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided